CLINICAL TRIAL: NCT04391257
Title: A Prospective Trial to Determine if it is Safe to Use the gekoTM Neuromuscular Electrostimulation Device in a Pacemaker Population.
Brief Title: Study of gekoTM Interaction With Cardiac Pacemakers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firstkind Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: FSK-CVD-003
Record Dates: First submitted 2020-04-30; First posted 2020-05-18 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Stroke; Wound Heal; Edema Leg; Cardiac Pacemaker Electrical Interference
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main (Other): gekoTM neuromuscular electrostimulation device (NMES) briefly used on patients with cardiac pacemakers to check if pacemakers detect the gekoTM electrical pulses as interference.
  Interventions: Device: geko™

INTERVENTIONS:
Device: geko™ — Assess if cardiac pacemakers detect geko™ electrical output pulse.

SUMMARY:
The gekoTM device is a small disposable battery powered device that attaches to the lower leg near the knee and stimulates the common peroneal nerve, causing muscle contraction of the lower leg. This contraction increases blood flow and the device is used to treat several conditions including deep vein thrombosis and venous leg ulcers.

There is evidence that some powered muscle stimulators and related devices can affect Cardiac Demand Pacemakers. This study is to ascertain if there is any such interaction between the gekoTM device and permanently implanted cardiac pacemakers.

DETAILED DESCRIPTION:
CFR.890.5850 requires that the labelling for powered muscle stimulators includes the contraindication 'Powered muscle stimulators should not be used on patients with cardiac demand pacemakers'.

Further, IEC 60601-2-10:2012 clause 210.7.9.2.101d, requires that the instructions for use provide: 'Advice that a PATIENT with an implanted electronic device (for example a cardiac pacemaker) should not be subjected to stimulation unless specialist medical opinion has first been obtained'. However, no details on what criteria the specialist should apply.

There is evidence that some powered muscle stimulators, and related devices can affect Cardiac Demand Pacemakers(1,2). Traditional powered muscle stimulators use pulse trains at a frequency of at least 30Hz(3) to elicit muscle contractions. The electrodes for these devices may be placed at number of sites on the body depending on the application, including the legs, arms and torso, often with well-spaced electrodes that may be attached to different limbs, sending electrical impulses through the torso.

The geko™ range of devices, however operate by delivering a single pulse at a frequency of 1Hz with electrodes placed topically, close together, at the knee. The nature of the stimulation pulse, and its location make it extremely unlikely that the geko™ devices could interfere with cardiac demand pacemakers. However, there is no direct evidence to support this assumption. This trial will determine if there are any adverse interactions between the geko™ and cardiac pacemakers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years and able to provide written informed consent.
* Intact healthy skin at the site of geko™ device application.
* Patient has a single, dual or bi-ventricular pacemaker implanted and is not pacing dependent.
* Patient understands and is willing to participate in the study and is able to comply with study procedures and visits.

Exclusion Criteria:

* Pregnancy or breast feeding.
* Use of any concurrent use of a neuro-modulation device.
* Any medication deemed by the Investigator to potentially interfere with the study treatment (e.g. systemic steroids.)
* Participation in any other clinical study that may interfere with the outcome of either study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is percentage of pacemaker sensed geko™ pulses in a 30 second period. | One day - single follow-up.
  Interference with pacemaker function.

SECONDARY OUTCOMES:
The secondary endpoints are the incidence of adverse events (AEs), incidence of serious AEs (SAEs), incidence of study treatment related AEs, and the incidence of investigational device related AEs. | One day-single follow-up.
  Incidence of adverse and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Zaheer Yousef, MD, Principal Investigator — University Hospital of Wales, Cardiff
Locations (2):
- United Kingdom (2):
  - University Hospital of Wales, Cardiff
  - The Dudley Group NHS Foundation Trust, Dudley